CLINICAL TRIAL: NCT03155945
Title: A Randomized, Open-label, Parallel, Phase 2a Study to Determine the Tolerability, Pharmacokinetics, and Efficacy of APD371 in Participants With Crohn's Disease Experiencing Abdominal Pain
Brief Title: Tolerability, Pharmacokinetics, and Efficacy of APD371 in Participants With Crohn's Disease Experiencing Abdominal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APD371-004
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Crohn's Disease; Abdominal Pain
MeSH Terms: conditions — Crohn Disease; Abdominal Pain | interventions — olorinab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olorinab 25 mg TID (Experimental): Participants received olorinab 25 milligrams (mg) tablet by mouth, three times daily (TID) for 8 weeks
  Interventions: Drug: Olorinab
- Olorinab 100 mg TID (Experimental): Participants received olorinab 100 mg oral tablets TID for 8 weeks
  Interventions: Drug: Olorinab

INTERVENTIONS:
Drug: Olorinab — Olorinab active treatment for 8 weeks.
  Other Names: APD371

SUMMARY:
The purpose of this randomized, open-label, parallel, phase 2a study is to determine the tolerability, pharmacokinetics, and efficacy of olorinab in participants with Crohn's disease experiencing abdominal pain.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of Crohn's disease for at least 3 months prior to screening corroborated by prior endoscopic and histopathologic documentation consistent with Crohn's disease.
* Quiescent to mildly active inflammatory Crohn's disease defined with a total of simple endoscopy score for Crohn's disease (SES-CD) score of < 10 or fecal calprotectin < 500 mcg/g within 4 weeks before Screening.
* Moderate to severe abdominal pain as defined by average abdominal pain score (AAPS) of >/= 4points on 7 consecutive days of the screening period up to Day -2. AAPS will be based on the 11-point numeric rating scale where 0 (no abdominal pain) to 10 (worst possible abdominal pain).

Key Exclusion Criteria:

* Female participants who are lactating or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 prior to study drug administration.
* Recent history (within 6 months of screening visit) of cerebrovascular disease, Acute Coronary Syndrome, Cerebrovascular accident, Transient ischemic attack, Myocardial infarction, unstable angina.
* Other significant chronic pain conditions that in the opinion of the Investigator may influence the abdominal pain score.
* History of extensive colonic resection, subtotal or total colectomy.
* History of >3 small bowel resections or diagnosis of short bowel syndrome or who have undergone bowel resection within 6 months prior to randomization.
* Chronic active hepatitis B within the last year (unless shown at the time of study entry to be hepatitis B antigen negative) or any history of hepatitis C.
* Evidence of current gastro-intestinal infection (bacterial or parasitic) or significant infection within 45 days of screening.

Note: other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (7):
- United States (7):
  - Clinical Research of Brandon, Brandon, Florida
  - Northwestern University, Chicago, Illinois
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Hassman Research Institute, Berlin, New Jersey
  - Wake Research Associates, Raleigh, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

REFERENCES:
- [Derived] Castro J, Garcia-Caraballo S, Maddern J, Schober G, Lumsden A, Harrington A, Schmiel S, Lindstrom B, Adams J, Brierley SM. Olorinab (APD371), a peripherally acting, highly selective, full agonist of the cannabinoid receptor 2, reduces colitis-induced acute and chronic visceral hypersensitivity in rodents. Pain. 2022 Jan 1;163(1):e72-e86. doi: 10.1097/j.pain.0000000000002314. PMID 33863856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were screened for the study. Of these, 23 participants failed screening, and 14 participants were randomized in the study.
Groups:
- Olorinab 100 mg TID: Participants received olorinab 100 mg tablet by mouth, TID for 8 weeks
Period: Overall Study
Arm/Group | Olorinab 25 mg TID | Olorinab 100 mg TID
Started | 6 | 8
Completed | 6 | 5
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other Reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized participants who received at least 1 dose of olorinab.
Groups:
- Olorinab 25 mg TID: Participants received olorinab 25 mg tablet by mouth, TID for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Olorinab 25 mg TID | Olorinab 100 mg TID | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.0 (10.81) | 36.9 (15.20) | 36.1 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was defined as an adverse event (AE) that occurred after first dose of olorinab. A SAE was any untoward medical occurrence that at any dose resulted in the following outcomes: death, was life-threatening, required/prolonged hospitalization, disability/incapacity, congenital anomaly/birth defect, and important medical events. Safety was assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.
Time Frame: Up to approximately 12 weeks
Population: Safety Population: All randomized participants who received at least 1 dose of olorinab.
Measure: Count of Participants; unit: Participants
Arm/Group | Olorinab 25 mg TID | Olorinab 100 mg TID
Number analyzed (Participants) | 6 | 8
Participants
  TEAEs | 4 | 6
  SAEs | 0 | 1

2. Other Pre Specified Outcome: Exploratory - Geometric Mean Maximum Observed Plasma Concentration (Cmax) of Olorinab and Its Metabolites at Week 8
Description: The result for this exploratory endpoint was not reported.
Time Frame: Week 8: Pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Exploratory - Median Time for Cmax (Tmax) of Olorinab and Its Metabolites at Week 8
Description: The result for this exploratory endpoint was not reported.
Time Frame: Week 8: Pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Exploratory - Mean Area Under the Concentration Time Curve From Time of Dosing to 8 Hours Post-dose (AUC0-8) of Olorinab and Its Metabolites at Week 8
Description: The result for this exploratory endpoint was not reported.
Time Frame: Week 0 (Day 1, Day 2), Week 8 (Day -1), Week 8: Pre-dose, 0.5, 1, 2, 4, 6 and 8 hours post-dose
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Exploratory - Mean Change in Abdominal Pain Score (APS) From Trough to Peak at Week 8
Description: The result for this exploratory endpoint was not reported.
Time Frame: Baseline; Week 8
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Exploratory - Change From Baseline in Average APS (AAPS)
Description: The result for this exploratory endpoint was not reported.
Time Frame: Baseline; Week 1, 2, 4, 6 and 8
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Exploratory - Number of Participants Who Were End-of-treatment Responders
Description: The result for this exploratory endpoint was not reported.
Time Frame: Week 8
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Exploratory - Number of Participants Who Were Weekly Responders
Description: The result for this exploratory endpoint was not reported.
Time Frame: Weeks 1, 2, 4, 6, and 8
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory - Number of Pain-free Days Per Week
Description: The result for this exploratory endpoint was not reported.
Time Frame: Week 1, Week 2, Week 4, Week 6, Week 8, and end of treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory - Number of Participants Who Used Pain Rescue Medication
Description: The result for this exploratory endpoint was not reported.
Time Frame: Up to Week 8
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory - Change From Baseline in C-reactive Protein (CRP) Levels at Week 4 and Week 8
Description: The result for this exploratory endpoint was not reported.
Time Frame: Baseline, Week 4, Week 8
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory - Change From Baseline in Fecal Calprotectin Levels at Week 4 and Week 8
Description: The result for this exploratory endpoint was not reported.
Time Frame: Baseline, Week 4, Week 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 12 weeks
Description: TEAE was defined as an adverse event (AE) that occurred after first dose of olorinab. A SAE was any untoward medical occurrence that at any dose resulted in the following outcomes: death, was life-threatening, required/prolonged hospitalization, disability/incapacity, congenital anomaly/birth defect, and important medical events.
Groups:
- Olorinab 25 mg TID: Participants received olorinab 25 milligrams (mg) oral tablets three times daily (TID) for 8 weeks
Arm/Group | Olorinab 25 mg TID | Olorinab 100 mg TID
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/8
Other Adverse Events (participants affected / at risk) | 4/6 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olorinab 25 mg TID (N=6) | Olorinab 100 mg TID (N=8)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olorinab 25 mg TID (N=6) | Olorinab 100 mg TID (N=8)
Conjunctivitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Injection site extravasation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 1
C-reactive protein decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03155945/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT03155945/SAP_001.pdf